CLINICAL TRIAL: NCT04043455
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Parallel-Group Study to Evaluate the Safety, Tolerability, and Efficacy of Olorinab in Subjects With Irritable Bowel Syndrome Experiencing Abdominal Pain
Brief Title: Olorinab in Irritable Bowel Syndrome With Predominant Constipation (IBS-C) and Irritable Bowel Syndrome With Predominant Diarrhea (IBS-D)
Acronym: CAPTIVATE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APD371-202
Record Dates: First submitted 2019-08-01; First posted 2019-08-02 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2022-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: Abdominal pain; Olorinab; APD371; Irritable bowel syndrome (IBS); IBS-C (IBS with predominant constipation); IBS-D (IBS with predominant diarrhea)
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain | interventions — olorinab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Olorinab low dose (Main Study) (Experimental)
  Interventions: Drug: Olorinab
- Olorinab medium dose (Main Study) (Experimental)
  Interventions: Drug: Olorinab
- Olorinab high dose (Main Study) (Experimental)
  Interventions: Drug: Olorinab
- Placebo (Main Study) (Placebo Comparator)
  Interventions: Drug: Placebo
- Olorinab (Long-Term Extension) (Experimental): Participants will receive olorinab based on their treatment assignment in the Main Study.
  Interventions: Drug: Olorinab

INTERVENTIONS:
Drug: Olorinab — Olorinab Dose 1 capsule or tablet by mouth, 3 times per day up to 12 weeks
  Other Names: APD371
  Arms: Olorinab low dose (Main Study)
Drug: Olorinab — Olorinab Dose 2 capsule or tablet by mouth, 3 times per day up to 12 weeks
  Other Names: APD371
  Arms: Olorinab medium dose (Main Study)
Drug: Olorinab — Olorinab Dose 3 capsule or tablet by mouth, 3 times per day up to 12 weeks
  Other Names: APD371
  Arms: Olorinab high dose (Main Study)
Drug: Placebo — Olorinab matching placebo capsule or tablet by mouth, 3 times per day up to 12 weeks
  Arms: Placebo (Main Study)
Drug: Olorinab — Olorinab Dose 2 capsule or tablet by mouth, 3 times per day up to 52 weeks
  Other Names: APD371
  Arms: Olorinab (Long-Term Extension)
Drug: Olorinab — Olorinab Dose 3 capsule or tablet by mouth, 3 times per day up to 52 weeks
  Other Names: APD371
  Arms: Olorinab (Long-Term Extension)

SUMMARY:
The purpose of this study is to determine whether olorinab is a safe and effective treatment for abdominal pain in participants with irritable bowel syndrome (IBS).

ELIGIBILITY:
Main Study Inclusion Criteria:

* Diagnosis of irritable bowel syndrome (IBS) with predominant constipation (IBS-C) or predominant diarrhea (IBS-D) according to Rome IV criteria at Visit 1 (Screening)
* Per the Rome IV diagnostic algorithm for IBS, participants 50 years of age and over are to have had one of the following with a result that rules out causes of abdominal pain other than IBS:

  1. Colonoscopy (within 10 years of Visit 1 [Screening])
  2. Flexible sigmoidoscopy and double contrast barium enema (within 5 years of Visit 1 [Screening])
  3. Computed tomography colonography (within 5 years of Visit 1 [Screening])

Main Study Exclusion Criteria:

* Diagnosis of IBS with mixed bowel habits (IBS-M) or unsubtyped IBS (IBS-U)
* Clinically relevant changes in dietary, lifestyle, or exercise regimen within 30 days prior to Visit 1 (Screening) that may confound efficacy assessments in the clinical judgment of the Investigator (or designee)
* Any colonic or major abdominal surgery (eg, bariatric surgery [including gastric banding], stomach surgery, small/large bowel surgery, or abdominal large vessel surgery). History of cholecystectomy is exclusionary for participants with IBS-D. For participants with IBS-C, a history of cholecystectomy more than 6 months prior to Visit 1 (Screening) is allowed. Procedures such as appendectomy, hysterectomy, caesarean section, or polypectomy are allowed as long as they have occurred at least 3 months prior to Visit 1 (Screening).

Long-Term Extension Inclusion Criteria:

•All participants must have completed the Main Study (including both Visit 8 [Week 12] and Visit 9 [Week 14])

Long-Term Extension Exclusion Criteria:

* Participant meets any exclusion criteria from the Main Study at the time of assessing eligibility for the LTE, unless approved by the Sponsor in advance.
* Participant had less than 75% overall compliance with eDiary entries during the Main Study.
* Participant deviated from the prescribed dosage regimen during the Main Study (ie, overall study treatment compliance less than 85% or more than 115%), unless approved by the Sponsor in advance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arena CT.gov Administrator, Study Director — Arena Pharmaceuticals
Locations (69):
- United States (69):
  - Accel Research Sites - Birmingham Clinical Research Unit, Birmingham, Alabama
  - Clinical Research Associates, LLC, Huntsville, Alabama
  - East Valley Gastroenterology and Hepatology Associates, Chandler, Arizona
  - Gilbert Center for Family Medicine, Gilbert, Arizona
  - Alliance Research Institute, Canoga Park, California
  - GW Research, Inc., Chula Vista, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - TriWest Research Associates, LLC, El Cajon, California
  - Diagnamics Inc., Encinitas, California
  - Prime Care Clinical Research, Laguna Hills, California
  - Om Research, Attn: Heather Blunt, Lancaster, California
  - San Diego Gastroenterology Medical Associates (CTNx), San Diego, California
  - Precision Research Institute, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - Advanced Rx Clinical Research Group, Inc., Westminster, California
  - Lynn Institute of Denver, Aurora, Colorado
  - Clinical Research of Brandon, LLC, Brandon, Florida
  - Qps Mra, Llc, South Miami, Florida
  - Precision Clinical Research, LLC., Sunrise, Florida
  - Presicion Research Center Inc, Tampa, Florida
  - Agile Clinical Research Trials LLC, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Gastroenterology Associates of Gainesville Georgia, Gainesville, Georgia
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Advanced Clinical Research, Attn to: Owen Havey, Meridian, Idaho
  - Claude Mandel Medical Center, Chicago, Illinois
  - Lemah Creek Clinical Research, Oakbrook Terrace, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - WestGlenGI, Shawnee Mission, Kansas
  - CroNOLA, LLC, Houma, Louisiana
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Frederick Gastroenterology Associates, Frederick, Maryland
  - Flint Clinical Research, PLLC, Flint, Michigan
  - Center for Pharmaceutical Research, LLC an AMR company, Kansas City, Missouri
  - Hassman Research Institute, Berlin, New Jersey
  - Long Island Gastrointestinal Research Group LLP, Great Neck, New York
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - Peters Medical Research, LLC, High Point, North Carolina
  - M3 Wake Research, Raleigh, North Carolina
  - Great Lakes Medical Research, Beachwood, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Family Practice Center of Wadsworth, Inc. dba New Venture Medical Research, Wadsworth, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Digestive Disease Specialists, Inc., Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Lynn Institute of Tulsa, Tulsa, Oklahoma
  - Oregon Center for Clinical Investigations, Inc. (OCCI, Inc.), Salem, Oregon
  - Susquehanna Research Group, LLC, Harrisburg, Pennsylvania
  - Care Access Research, Pottsville, Pottsville, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Meridian Clinical Research, LLC, Dakota Dunes, South Dakota
  - Chattanooga Research & Medicine, PLLC, Chattanooga, Tennessee
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Biopharma Informatic, LLC, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Research Studies at Fine Digestive Health, Irving, Texas
  - ACR Gut Whisperer, West Jordan, Utah
  - New River Valley Research Institute, Christiansburg, Virginia
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
  - Exemplar Research Inc, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang L, Cash BD, Lembo A, Kunkel DC, English BA, Lindstrom B, Gu G, Skare S, Gilder K, Turner S, Cataldi F, Lipkis D, Tack J. Efficacy and safety of olorinab, a full agonist of the cannabinoid receptor 2, for the treatment of abdominal pain in patients with irritable bowel syndrome: Results from a phase 2b randomized placebo-controlled trial (CAPTIVATE). Neurogastroenterol Motil. 2023 May;35(5):e14539. doi: 10.1111/nmo.14539. Epub 2023 Feb 5. PMID 36740814

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-treatment period study (12-week Main Study Double-Blind Treatment Period and 52-week Double-Blind Long-Term Extension [LTE] Treatment Period) to assess the efficacy, safety and tolerability of Olorinab in the treatment of abdominal pain in participants with irritable bowel syndrome (IBS), who were not on concomitant treatment for IBS.
Pre-assignment Details: A total of 273 participants were enrolled into the 12-week Main Study Period and a total of 105 participants continued into the 52-week LTE Period.
Groups:
- Main Study Period: Olorinab 10 mg: Participants were randomized to receive Olorinab 10 mg 3 times per day (TID) for 12 Weeks. After completion of the Main Study, participants in this arm could continue to the LTE Period and were re-randomized to receive either 25 mg or 50 mg Olorinab.
- Main Study Period: Olorinab 25 mg: Participants were randomized to receive Olorinab 25 mg TID for 12 Weeks. After completion of the Main Study, participants in this arm could continue to receive the same dose in the LTE Period.
- Main Study Period: Olorinab 50 mg: Participants were randomized to receive Olorinab 50 mg TID for 12 Weeks. After completion of the Main Study, participants in this arm could continue to receive the same dose in the LTE Period.
- Main Study Period: Placebo: Participants were randomized to receive placebo TID for 12 Weeks. After completion of the Main Study, participants in this arm could continue to the LTE Period and were re-randomized to receive either 25 mg or 50 mg Olorinab.
- LTE Period: Olorinab 25 mg: Participants who successfully completed 12 weeks of treatment in the Main Study received Olorinab 25 mg TID for 52 weeks. During the Main study, participants in this arm had received Olorinab 25 mg or had received Olorinab 10 mg or placebo and were then re-randomized to the 25 mg dose for the LTE Period.
- LTE Period: Olorinab 50 mg: Participants who successfully completed 12 weeks of treatment in the Main Study received Olorinab 50 mg TID for 52 weeks. During the Main study, participants in this arm had received Olorinab 50 mg or had received Olorinab 10 mg or placebo and were then re-randomized to the 50 mg dose for the LTE Period.
Period: Main Study Double-Blind Treatment Period
Arm/Group | Main Study Period: Olorinab 10 mg | Main Study Period: Olorinab 25 mg | Main Study Period: Olorinab 50 mg | Main Study Period: Placebo | LTE Period: Olorinab 25 mg | LTE Period: Olorinab 50 mg
Started | 67 | 67 | 69 | 70 | 0 | 0
Received Treatment | 67 | 66 | 69 | 70 | 0 | 0
Completed | 59 | 53 | 61 | 58 | 0 | 0
Not Completed | 8 | 14 | 8 | 12 | 0 | 0
Not completed — Adverse Event | 2 | 3 | 2 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 4 | 9 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Regional site closure order due to Covid 19 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Did not receive treatment | 0 | 1 | 0 | 0 | 0 | 0
Period: Double-Blind LTE Treatment Period
Arm/Group | Main Study Period: Olorinab 10 mg | Main Study Period: Olorinab 25 mg | Main Study Period: Olorinab 50 mg | Main Study Period: Placebo | LTE Period: Olorinab 25 mg | LTE Period: Olorinab 50 mg
Started | 0 | 0 | 0 | 0 | 53 | 52
Received Treatment | 0 | 0 | 0 | 0 | 53 | 51
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 53 | 52
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 5 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Study termination by Sponsor | 0 | 0 | 0 | 0 | 47 | 44

BASELINE CHARACTERISTICS:
Population: Full Analysis Set comprises of all randomized participants irrespective of whether they received study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study Period: Olorinab 10 mg | Main Study Period: Olorinab 25 mg | Main Study Period: Olorinab 50 mg | Main Study Period: Placebo | Total
Number analyzed (Participants) | 67 | 67 | 69 | 70 | 273
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.5 (11.47) | 39.0 (12.68) | 39.5 (12.98) | 41.8 (14.38) | 40.4 (12.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 49 | 50 | 49 | 197
  Male | 18 | 18 | 19 | 21 | 76
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 0 | 3
  Asian | 2 | 5 | 10 | 5 | 22
  Black or African American | 22 | 12 | 17 | 14 | 65
  Multiple races | 0 | 1 | 0 | 0 | 1
  White | 38 | 46 | 39 | 50 | 173
  Not reported | 4 | 1 | 3 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Change From Baseline in Average Abdominal Pain Score (AAPS) at Week 12
Description: The APS is a single question, 11-point numeric rating scale in which 0 represents no abdominal pain and 10 represents the worst possible abdominal pain. The change in AAPS from Baseline at Week 12 was analyzed using a mixed-effects model repeated measures (MMRM) analysis with treatment, stratification factors, week, and treatment-by-week interaction as factors and Baseline AAPS as a covariate. An unstructured variance-covariance matrix was used for the MMRM analysis.
Time Frame: Baseline and Week 12
Population: Main Study Full Analysis Set. Only those participants with data available at the specified timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Groups:
- Main Study Period: Olorinab 10 mg: Participants were randomized to receive Olorinab 10 mg TID for 12 Weeks.
- Main Study Period: Olorinab 25 mg: Participants were randomized to receive Olorinab 25 mg TID for 12 Weeks.
- Main Study Period: Olorinab 50 mg: Participants were randomized to receive Olorinab 50 mg TID for 12 Weeks.
- Main Study Period: Placebo: Participants were randomized to receive placebo TID for 12 Weeks.
Arm/Group | Main Study Period: Olorinab 10 mg | Main Study Period: Olorinab 25 mg | Main Study Period: Olorinab 50 mg | Main Study Period: Placebo
Number analyzed (Participants) | 49 | 46 | 55 | 52
Scores on a scale | -2.32 (0.293) | -2.45 (0.297) | -2.68 (0.285) | -2.14 (0.289)
Statistical Analysis 1: Comparison: Main Study Period: Olorinab 10 mg vs Main Study Period: Placebo; Treatment comparison between Olorinab 10 mg and placebo using least square mean difference and 95% confidence interval (CI) has been presented; Test type: Superiority; p = 0.650, Mixed Models Analysis; Least square mean difference = -0.19, 95% CI 2-sided [-0.99 to 0.62], Standard Error of Mean 0.407
Statistical Analysis 2: Comparison: Main Study Period: Olorinab 25 mg vs Main Study Period: Placebo; Treatment comparison between Olorinab 25 mg and placebo using least square mean difference and 95% CI has been presented; Test type: Superiority; p = 0.439, Mixed Models Analysis; Least square mean difference = -0.32, 95% CI 2-sided [-1.12 to 0.49], Standard Error of Mean 0.409
Statistical Analysis 3: Comparison: Main Study Period: Olorinab 50 mg vs Main Study Period: Placebo; Treatment comparison between Olorinab 50 mg and placebo using least square mean difference and 95% CI has been presented; Test type: Superiority; p = 0.172, Mixed Models Analysis; Least square mean difference = -0.55, 95% CI 2-sided [-1.34 to 0.24], Standard Error of Mean 0.401

2. Primary Outcome: Main Study: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a medicinal product without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were defined as any AE that started or worsened in severity on or after the first dose of study treatment.
Time Frame: Up to 14 Weeks
Population: Main Study Safety Set comprises of participants randomly assigned to study treatment and who took at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Period: Olorinab 10 mg | Main Study Period: Olorinab 25 mg | Main Study Period: Olorinab 50 mg | Main Study Period: Placebo
Number analyzed (Participants) | 67 | 66 | 69 | 70
Participants
  Any TEAEs | 34 | 33 | 31 | 35
  Any SAEs | 0 | 0 | 0 | 0

3. Primary Outcome: LTE Period: Number of Participants With TEAEs and SAEs
Description: An AE was any untoward medical occurrence in a participant administered a medicinal product without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were defined as any AE that started or worsened in severity on or after the first dose of study treatment.
Time Frame: Up to 54 Weeks
Population: LTE Period Safety Set comprises of participants randomly assigned to study treatment and who took at least one dose of study treatment in the LTE Period.
Measure: Count of Participants; unit: Participants
Arm/Group | LTE Period: Olorinab 25 mg | LTE Period: Olorinab 50 mg
Number analyzed (Participants) | 53 | 51
Participants
  Any TEAEs | 17 | 14
  Any SAEs | 0 | 0

4. Primary Outcome: Main Study: Number of Participants With Clinically Significant Abnormal Laboratory Parameters
Description: Blood samples were collected for the analysis of laboratory parameters including serum chemistry, hematology, coagulation, and urinalysis. The investigator was responsible for reviewing laboratory results for clinically significant abnormalities.
Time Frame: Baseline to Week 14
Population: Main Study Safety Set.
Measure: Count of Participants; unit: Participants
Groups:
- Olorinab 10 mg: Participants in this arm received Olorinab 10 mg 3 times per day for 12 Weeks.
- Olorinab 25 mg: Participants in this arm received Olorinab 25 mg 3 times per day for 12 Weeks.
- Olorinab 50 mg: Participants in this arm received Olorinab 50 mg 3 times per day for 12 Weeks.
- Placebo: Participants in this arm received placebo 3 times per day for 12 Weeks.
Arm/Group | Olorinab 10 mg | Olorinab 25 mg | Olorinab 50 mg | Placebo
Number analyzed (Participants) | 67 | 66 | 69 | 70
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: LTE Study: Number of Participants With Clinically Significant Abnormal Laboratory Parameters
Description: as for outcome 4
Time Frame: Baseline to Week 54 (of LTE)
Population: LTE Safety Set.
Measure: Count of Participants; unit: Participants
Arm/Group | LTE Period: Olorinab 25 mg | LTE Period: Olorinab 50 mg
Number analyzed (Participants) | 53 | 51
Participants | 0 | 1

6. Primary Outcome: Main Study: Number of Participants With Clinically Significant Abnormal Vital Signs
Description: Parameters assessed for vital signs included blood pressure (systolic and diastolic blood pressure), heart rate (HR), body temperature, and respiratory rate. The investigator was responsible for reviewing vital signs for clinically significant abnormalities.
Time Frame: Baseline to Week 14
Population: Main Study Safety Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study Period: Olorinab 10 mg | Main Study Period: Olorinab 25 mg | Main Study Period: Olorinab 50 mg | Main Study Period: Placebo
Number analyzed (Participants) | 67 | 66 | 69 | 70
Participants | 0 | 0 | 0 | 0

7. Primary Outcome: LTE Study: Number of Participants With Clinically Significant Abnormal Vital Signs
Description: Parameters assessed for vital signs included blood pressure (systolic and diastolic blood pressure), HR, body temperature, and respiratory rate. The investigator was responsible for reviewing vital signs for clinically significant abnormalities.
Time Frame: Baseline to Week 54 (of LTE)
Population: LTE Safety Set.
Measure: Count of Participants; unit: Participants
Arm/Group | LTE Period: Olorinab 25 mg | LTE Period: Olorinab 50 mg
Number analyzed (Participants) | 53 | 51
Participants | 0 | 0

8. Secondary Outcome: Main Study: Percentage of Participants Achieving a Greater Than or Equal to (>=) 30% Improvement in AAPS at Week 12
Description: The percentage of participants achieving a >= 30% improvement in AAPS from Baseline at Week 12 was analyzed using a Cochran-Mantel-Haenszel (CMH) test stratified by the stratification factors. Missing post-baseline AAPS data was imputed using multiple imputation (MI) under the missing at random (MAR) assumption. Participants who were randomized but did not have at least 1 post-Baseline observation were considered non-responders. A >= 30% improvement in AAPS was a reduction in AAPS of 30% or more when compared to Baseline AAPS.
Time Frame: Baseline and Week 12
Population: Main Study Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study Period: Olorinab 10 mg | Main Study Period: Olorinab 25 mg | Main Study Period: Olorinab 50 mg | Main Study Period: Placebo
Number analyzed (Participants) | 67 | 67 | 69 | 70
Percentage of participants | 56.7 [44.85 to 68.58] | 59.7 [47.96 to 71.45] | 56.5 [44.82 to 68.22] | 52.9 [41.16 to 64.55]
Statistical Analysis 1: Comparison: Main Study Period: Olorinab 10 mg vs Main Study Period: Placebo; Treatment comparison between Olorinab 10 mg and placebo using Odds ratio and 95% CI has been presented; Test type: Superiority; p = 0.659, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.156, 95% CI 2-sided [-0.019 to 2.331]
Statistical Analysis 2: Comparison: Main Study Period: Olorinab 25 mg vs Main Study Period: Placebo; Treatment comparison between Olorinab 25 mg and placebo using Odds ratio and 95% CI has been presented; Test type: Superiority; p = 0.557, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.248, 95% CI 2-sided [-0.040 to 2.535]
Statistical Analysis 3: Comparison: Main Study Period: Olorinab 50 mg vs Main Study Period: Placebo; Treatment comparison between Olorinab 50 mg and placebo using Odds ratio and 95% CI has been presented; Test type: Superiority; p = 0.541, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.245, 95% CI 2-sided [0.027 to 2.462]

9. Secondary Outcome: Main Study: Percentage of Participants Achieving a >= 30% Improvement in AAPS From Baseline for at Least 6 of the 12 Weeks
Description: The percentage of participants achieving a >= 30% improvement in AAPS from Baseline for at least 6 of the 12 weeks during the Treatment Period were analyzed using a CMH test stratified by the stratification factors. A >= 30% improvement in AAPS is a reduction in AAPS of 30% or more when compared to Baseline AAPS. Missing post-baseline AAPS data was imputed using MI under the MAR assumption.
Time Frame: Baseline and Week 12
Population: Main Study Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study Period: Olorinab 10 mg | Main Study Period: Olorinab 25 mg | Main Study Period: Olorinab 50 mg | Main Study Period: Placebo
Number analyzed (Participants) | 67 | 67 | 69 | 70
Percentage of participants | 53.7 [41.79 to 65.67] | 53.7 [41.79 to 65.67] | 53.6 [41.86 to 65.39] | 47.1 [35.45 to 58.84]
Statistical Analysis 1: Comparison: Main Study Period: Olorinab 10 mg vs Main Study Period: Placebo; Treatment comparison between Olorinab 10 mg and placebo using Odd's ratio and 95% CI has been presented; Test type: Superiority; p = 0.529, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.234, 95% CI 2-sided [-0.001 to 2.468]
Statistical Analysis 2: Comparison: Main Study Period: Olorinab 25 mg vs Main Study Period: Placebo; Treatment comparison between Olorinab 25 mg and placebo using Odd's ratio and 95% CI has been presented; Test type: Superiority; p = 0.730, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.123, 95% CI 2-sided [0.015 to 2.232]
Statistical Analysis 3: Comparison: Main Study Period: Olorinab 50 mg vs Main Study Period: Placebo; Treatment comparison between Olorinab 50 mg and placebo using Odd's ratio and 95% CI has been presented; Test type: Superiority; p = 0.548, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.226, 95% CI 2-sided [0.025 to 2.428]

10. Secondary Outcome: Main Study: Percent Change From Baseline in AAPS at Week 12
Description: The percent change in AAPS from Baseline at Week 12 was analyzed using an MMRM analysis with treatment, stratification factors, week, and treatment-by-week interaction as factors and Baseline AAPS as a covariate. Baseline is the last non-missing measurement collected prior to the first dose of study treatment at Day 1.
Time Frame: Baseline and Week 12
Population: Main Study Full Analysis Set. Only those participants with data available at the specified timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Main Study Period: Olorinab 10 mg | Main Study Period: Olorinab 25 mg | Main Study Period: Olorinab 50 mg | Main Study Period: Placebo
Number analyzed (Participants) | 49 | 46 | 55 | 52
Percent change | -36.91 (4.459) | -37.73 (4.521) | -38.44 (4.327) | -34.48 (4.388)
Statistical Analysis 1: Comparison: Main Study Period: Olorinab 10 mg vs Main Study Period: Placebo; Treatment comparison between Olorinab 10 mg and placebo using least square mean difference and 95% CI has been presented; Test type: Superiority; p = 0.696, Mixed Models Analysis; Least square mean difference = -2.42, 95% CI 2-sided [-14.61 to 9.76], Standard Error of Mean 6.189
Statistical Analysis 2: Comparison: Main Study Period: Olorinab 25 mg vs Main Study Period: Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.602, Mixed Models Analysis; Least square mean difference = -3.25, 95% CI 2-sided [-15.51 to 9.00], Standard Error of Mean 6.222
Statistical Analysis 3: Comparison: Main Study Period: Olorinab 50 mg vs Main Study Period: Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.516, Mixed Models Analysis; Least square mean difference = -3.96, 95% CI 2-sided [-15.95 to 8.03], Standard Error of Mean 6.088

11. Secondary Outcome: Main Study: Change From Baseline in Number of Pain-Free Days at Week 12
Description: The change from Baseline at Week 12 in number of pain-free days per week was analyzed using a MMRM analysis with treatment, stratification factors, week, and treatment-by-week interaction as factors and Baseline pain free days as a covariate. Pain-free days were defined as days with a pain score of zero (0). Baseline is the last non-missing measurement collected prior to the first dose of study treatment at Day 1.
Time Frame: Baseline and Week 12
Population: Main Study Full Analysis Set. Only those participants with data available at the specified timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Days per week
Arm/Group | Main Study Period: Olorinab 10 mg | Main Study Period: Olorinab 25 mg | Main Study Period: Olorinab 50 mg | Main Study Period: Placebo
Number analyzed (Participants) | 49 | 46 | 55 | 52
Days per week | 0.61 (0.218) | 0.39 (0.222) | 0.66 (0.213) | 0.54 (0.216)
Statistical Analysis 1: Comparison: Main Study Period: Olorinab 10 mg vs Main Study Period: Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.804, Mixed Models Analysis; Least square mean difference = 0.08, 95% CI 2-sided [-0.53 to 0.68], Standard Error of Mean 0.305
Statistical Analysis 2: Comparison: Main Study Period: Olorinab 25 mg vs Main Study Period: Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.618, Mixed Models Analysis; Least square mean difference = -0.15, 95% CI 2-sided [-0.76 to 0.45], Standard Error of Mean 0.308
Statistical Analysis 3: Comparison: Main Study Period: Olorinab 50 mg vs Main Study Period: Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.687, Mixed Models Analysis; Least square mean difference = 0.12, 95% CI 2-sided [-0.47 to 0.71], Standard Error of Mean 0.301

12. Secondary Outcome: Main Study: Maximum Concentration (Cmax) of Olorinab
Description: Blood samples were collected from participants at indicated timepoints after the administration of study treatment to investigate Cmax of Olorinab. Pharmacokinetic (PK) analysis was conducted using standard non-compartmental methods.
Time Frame: On Day 1: Pre-dose and 0.5, 1, 2, 4, and 8 hours post dose and Week 4: Pre-dose and 0.5, 1 and 2 hours post dose
Population: Main Study PK Analysis Set comprises of all participants in the Full Analysis Set with at least one post-dose PK parameter. Only those participants with data available at the specified timepoints were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Main Study Period: Olorinab 10 mg | Main Study Period: Olorinab 25 mg | Main Study Period: Olorinab 50 mg
Number analyzed (Participants) | 56 | 53 | 58
Nanograms per milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 24 | 24 | 22
  Day 1 | 296.4 (51.48) | 591.2 (57.16) | 963.7 (107.4)
  Week 4 | 320.5 (123.4) | 361.7 (350.4) | 1097 (113.4)

13. Secondary Outcome: Main Study: Time of Maximum Concentration After Drug Administration (Tmax) of Olorinab
Description: Blood samples were collected from participants at indicated timepoints after the administration of study treatment to investigate Tmax of Olorinab. PK analysis was conducted using standard non-compartmental methods.
Time Frame: On Day 1: Pre-dose and 0.5, 1, 2, 4, and 8 hours post dose and Week 4: Pre-dose and 0.5, 1 and 2 hours post dose
Population: Main Study PK Analysis Set. Only those participants with data available at the specified timepoints were analyzed. Sampling times reflected timeframe based on actual time and not planned nominal time.
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study Period: Olorinab 10 mg | Main Study Period: Olorinab 25 mg | Main Study Period: Olorinab 50 mg
Number analyzed (Participants) | 53 | 51 | 54
Hours
  Day 1: number analyzed (Participants) | 23 | 24 | 21
  Day 1 | 1.00 [1.00 to 4.27] | 2.02 [0.50 to 4.15] | 1.02 [0.50 to 8.08]
  Week 4 | 1.00 [0.00 to 2.25] | 1.00 [0.00 to 2.48] | 1.00 [0.00 to 2.05]

14. Secondary Outcome: Main Study: Plasma Trough Concentrations (Ctrough) of Olorinab
Description: Blood samples were collected from participants at indicated time frames after the administration of study treatment to investigate Ctrough of Olorinab. PK analysis was conducted using standard non-compartmental methods.
Time Frame: Pre dose on Day 1, Day 2 and Weeks 2, 4, 8, 10 and 12
Population: Main Study PK Analysis Set. Only those participants with data available at the specified timepoints were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Main Study Period: Olorinab 10 mg | Main Study Period: Olorinab 25 mg | Main Study Period: Olorinab 50 mg
Number analyzed (Participants) | 32 | 30 | 27
ng/mL
  Day 1: number analyzed (Participants) | 15 | 17 | 18
  Day 1 | 32.46 (166.4) | 88.07 (183.2) | 150.7 (130.1)
  Day 2: number analyzed (Participants) | 14 | 18 | 17
  Day 2 | 74.70 (85.04) | 244.7 (81.41) | 266.7 (174.7)
  Week 2: number analyzed (Participants) | 27 | 27 | 25
  Week 2 | 39.41 (255.6) | 109.8 (317.2) | 125.2 (233.3)
  Week 4 | 48.23 (323.8) | 77.71 (205.8) | 140.6 (320.0)
  Week 8: number analyzed (Participants) | 20 | 23 | 22
  Week 8 | 50.45 (146.9) | 111.4 (243.2) | 200.3 (180.4)
  Week 10: number analyzed (Participants) | 25 | 19 | 27
  Week 10 | 32.69 (296.8) | 45.96 (470.8) | 137.3 (1193)
  Week 12: number analyzed (Participants) | 18 | 20 | 20
  Week 12 | 50.39 (136.8) | 84.09 (471.9) | 102.0 (288.4)

ADVERSE EVENTS:
Time Frame: TEAEs and SAEs were collected from Day 1 up to Week 14 of the Main Study Treatment Period and from Day 1 up to Week 54 of the LTE Period.
Description: TEAEs and SAEs were collected in the Safety Set which comprised of participants randomly assigned to study treatment and who took at least one dose of study treatment in the Main Study Period or LTE Period, as applicable.
Arm/Group | Main Study Period: Olorinab 10 mg | Main Study Period: Olorinab 25 mg | Main Study Period: Olorinab 50 mg | Main Study Period: Placebo | LTE Period: Olorinab 25 mg | LTE Period: Olorinab 50 mg
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/66 | 0/69 | 0/70 | 0/53 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/66 | 0/69 | 0/70 | 0/53 | 0/51
Other Adverse Events (participants affected / at risk) | 34/67 | 33/66 | 31/69 | 35/70 | 17/53 | 14/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study Period: Olorinab 10 mg (N=67) | Main Study Period: Olorinab 25 mg (N=66) | Main Study Period: Olorinab 50 mg (N=69) | Main Study Period: Placebo (N=70) | LTE Period: Olorinab 25 mg (N=53) | LTE Period: Olorinab 50 mg (N=51)
Nasopharyngitis (Infections and infestations) | 5 | 1 | 3 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 5 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 4 | 1 | 1
Bacterial vaginosis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 3 | 5 | 1 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 3 | 1 | 2 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 1
Headache (Nervous system disorders) | 6 | 2 | 3 | 2 | 0 | 3
Dizziness (Nervous system disorders) | 4 | 1 | 2 | 1 | 1 | 1
Somnolence (Nervous system disorders) | 3 | 0 | 3 | 0 | 0 | 0
Migraine (Nervous system disorders) | 2 | 1 | 0 | 2 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 1
Drug withdrawal headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Orthostatic intolerance (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 2 | 2 | 0 | 0 | 0
Protein urine present (Investigations) | 1 | 2 | 1 | 0 | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 2 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 1 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 2 | 1 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 2 | 0
Blood pressure increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 0
Nitrite urine present (Investigations) | 0 | 2 | 0 | 0 | 1 | 0
Urine bilirubin increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 1
Urine ketone body present (Investigations) | 0 | 2 | 0 | 0 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 1 | 1 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
SARS-COV-2 test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
White blood cells urine positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram PR prolongation (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 1 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 2 | 1
Bilirubinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 2 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Medical device site irritation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Multiple allergies (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lice Infestation (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Onchomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic Steotosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT04043455/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT04043455/SAP_001.pdf